CLINICAL TRIAL: NCT05506826
Title: Effects of Mirror Therapy Versus Fine Motor Activities on Hand Function in Chronic Stroke Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/21/0254
Record Dates: First submitted 2022-08-17; First posted 2022-08-18 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Stroke, Ischemic; Acute Pain; Weakness, Muscle
Keywords: Stroke, Ischemic; Acute Pain; Weakness, Muscle
MeSH Terms: conditions — Ischemic Stroke; Acute Pain; Muscle Weakness | interventions — Mirror Movement Therapy

STUDY DESIGN:
Intervention Model Description: Study participants will be divided in two groups. Patients in group A will receive conventional therapy for four weeks sixty minutes per day, five days per week. In Group B patients will perform fine motor exercises like therapy ball exercises, therapy putty exercises, table top exercises, moving beans, stacking pennies and rubber band resistances exercises etc. for 30 minutes along with conventional therapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fine motor activities group (Experimental): Patients in this group will receive conventional therapy for 1 month sixty minutes/day, 5 days/week in addition to performing fine motor exercises like therapy ball exercises, therapy putty exercises, table top exercises, moving beans, stacking pennies and rubber band resistances exercises etc. for 30 minutes
  Interventions: Other: fine motor activities
- control group (Active Comparator): Patients in this group will receive conventional therapy for four weeks sixty minutes per day, five days per week. In addition, receive thirty minutes of mirror therapy, which included periodic wrist flexion-extension, flexion and extension exercises of fingers on non paralyzed limb
  Interventions: Other: conventional therapy and mirror therapy

INTERVENTIONS:
Other: fine motor activities — patient will perform fine motor exercises like therapy ball exercises, therapy putty exercises, table top exercises, moving beans, stacking pennies and rubber band resistances exercises etc. for 30 minutes along with conventional therapy
  Arms: fine motor activities group
Other: conventional therapy and mirror therapy — Patients in this group will receive conventional therapy for four weeks sixty minutes per day, five days per week. In addition, receive thirty minutes of mirror therapy, which included periodic wrist flexion-extension, flexion and extension exercises of fingers on non paralyzed limb
  Arms: control group

SUMMARY:
to compare the effects of the Mirror therapy and fine motor activities on hand function in chronic stroke patients

DETAILED DESCRIPTION:
This study will be conducted to compare the effects of mirror therapy and fine motor activities in chronic stroke patients. Total Twenty eight hemiplegic patients will be recruited according to inclusion criteria and data will be collected from Riphah rehabilitation centre Lahore and Mian Munshi Hospital Lahore (DHQ). The patients will randomly assigned to a mirror therapy group (n=14) and Fine motor activities group (n=14). The patients in both groups will undergo conventional therapy for 4 weeks (60minutes/day, 5 days/week). The patients will be evaluated at the beginning and end of the treatment by Fugl- Meyer Aassessment (FMA) wolf motor assessment scale and the Functional Independence Measure (FIM). After approval from ethical committee, data collection will be started and informed consent will be taken from all patients.

ELIGIBILITY:
Inclusion Criteria:

* A score greater than 24 on the Mini-Mental State examination test
* Chronic stroke patients whose episode of stroke onset was 6 months to 2 years.
* Patients who are able to communicate well and grasp the therapist's spoken instructions

Exclusion Criteria:

* Patients who have restricted joint movement in their healthy upper extremities.
* Neglect syndrome or a visual field deficiency
* Patients with recurrent stroke.
* Spine surgery.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-08-20 (Actual); Study Completion 2022-08-20 (Actual)

PRIMARY OUTCOMES:
fugl mayer assessment FMA upper limb | 9 months
  For stroke patients, the Fugal-Meyer Assessment (FMA) is a performance-based impairment measure. It is used to assess balance, motor function, sensation, and joint function in persons who suffer hemiplegia after a stroke. In both clinical and research settings, it is used to identify sickness severity, define motor recovery, and plan and assess treatment
The Functional Independence Measure (FIM) | 9 months
  The Functional Independence Measure (FIM) is a non-diagnostic disability assessment instrument that was developed for a wide range of groups
The Wolf Motor Function Test (WMFT) | 9 months
  The Wolf Motor Function Test (WMFT) uses timed and functional tasks to assess upper limb motor skills

CONTACTS AND LOCATIONS:
Overall Officials: zeest hashmi, MSNMPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Fedral, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hillis AE. Developments in treating the nonmotor symptoms of stroke. Expert Rev Neurother. 2020 Jun;20(6):567-576. doi: 10.1080/14737175.2020.1763173. Epub 2020 May 12. PMID 32363957
- [Background] Gandhi DB, Sterba A, Khatter H, Pandian JD. Mirror Therapy in Stroke Rehabilitation: Current Perspectives. Ther Clin Risk Manag. 2020 Feb 7;16:75-85. doi: 10.2147/TCRM.S206883. eCollection 2020. PMID 32103968
- [Background] Umeki N, Murata J, Higashijima M. Effects of Training for Finger Perception on Functional Recovery of Hemiplegic Upper Limbs in Acute Stroke Patients. Occup Ther Int. 2019 Nov 4;2019:6508261. doi: 10.1155/2019/6508261. eCollection 2019. PMID 31777474
- [Background] Fong KNK, Ting KH, Chan CCH, Li LSW. Mirror therapy with bilateral arm training for hemiplegic upper extremity motor functions in patients with chronic stroke. Hong Kong Med J. 2019 Feb;25 Suppl 3(1):30-34. No abstract available. PMID 30792371